CLINICAL TRIAL: NCT05784272
Title: A Multi-centred Exploratory Study Investigating the Determinants of Progression From Phase III to Phase IV Cardiac Rehabilitation in Underrepresented Populations
Brief Title: Determinants of Progression From Phase III to IV Cardiac Rehabilitation
Status: Recruiting | Type: Observational
Sponsor: Manchester Metropolitan University (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Principal Investigator, Stefan Birkett, Senior Lecturer in Cardiovascular Rehabilitation, Manchester Metropolitan University
Other Study IDs: IRAS: 322092
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular; Rehabilitation; Underepresented groups
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Initiators: These will be the participants who initiate into phase IV cardiac reahb
- Non-initiators: These will be the participants who do not initiate into phase IV cardiac reahb

SUMMARY:
This study will determine the limiting factors in progression from phase III to IV cardiac rehabilitation in underepresented populations (as defined by the National Audit of Cardiac Rehab, NACR). This will be done by recruiting participants from phase III cardiac rehab programmes and issuing questionnaires (either a non-initiator questionnire, or an initiator questionnaire based on if the participant is intiating into phase IV cardiac rehab. The questionnaires will assess reasons for/against progression as well as collecting some demographic and data indicative of socioeconomic status. Semi-structured interviews will then be conducted to assess reasons/barriers for progression to phase IV in a convenience sample of both initiators and non-initiators.

DETAILED DESCRIPTION:
In the United Kingdom (UK) >2.3 million people are living with coronary heart disease (CHD) (1). Cardiac rehabilitation (CR) is a core component of secondary prevention that reduces hospitalisations, cardiovascular mortality and improves quality of life (2). Traditionally, CR has four phases: Phase I (in-hospital), Phase II (early outpatient), Phase III (early CR typically 8-11 weeks in duration) and Phase IV, the long-term maintenance programme which aims to further build on the success of Phase III (3). As longer-term CR programmes (beyond 11 weeks) are associated with reductions in mortality, greater gains in fitness and improvement in risk factors (4-6), it is important that patients are encouraged to continue to take part in CR for as long as possible. Despite the associated benefits of CR, pre-Covid-19, only 50% of those eligible in the UK accessed Phase III (7) with this percentage further decreasing during the pandemic to 36%. A major concern was that there was a further reduction of 11% and 6% in ethnic minorities and female participation, two groups already significantly underrepresented in CR (7). Consequently, the most recent National Audit of Cardiac Rehabilitation (NACR) report (2021) stated that the development and implementation of strategies to halt the widening gap is a key priority. Data regarding uptake for long-term phase IV CR are limited (8).

Patient Identification Patients who are currently attending a Phase III cardiac rehabilitation programme at the aforementioned centres and who meet the inclusion criteria will be approached by members of the cardiac rehabilitation team at each site. If patients agree verbal and written information will be provided.

Consent The phase III CR team from each centre will explain what participating in this study would involve and give them a participant information sheet. The potential participant will then be given the opportunity to ask the phase III staff member and questions they may have. If the phase III staff member is not sure, the research team will be contacted, and clarification will be provided. Only those capable of giving informed consent will be eligible to participate. This includes being able to understand and communicate in English language well enough to give informed consent as no translation will be available in this study. Verbal and written informed consent to partake in the study and to be contacted by the research team will be attained at the patients Phase III discharge assessment by a member of the cardiac rehabilitation team. Institutional email addresses will be used to inform the research team of patients who have given informed consent (NHS email addresses from the rehabilitation team sending to Manchester Metropolitan University email addresses of the research team). The informed consent documents will be scanned and emailed to the research team and then the physical copies will be destroyed at the Trust's site. The research team will then hold these documents in a password protected folder on Manchester Metropolitan University's secure dropbox system. In compliance with the Welsh Language Act 1993, where participant information sheets and informed consent forms will be translated into Welsh where this is requested by a participant.

Study procedures At least one week prior to their Phase III discharge assessment, eligible patient will be given a patient information sheet. They will have the opportunity to ask any questions relating to the study. At their final phase III assessment, they will be asked if they would like to participate and informed consent and consent to contact will be obtained. Consented CR participants will be contacted by the research team and asked to complete a digital or paper form questionnaire based on their choice to initiate or not to initiate Phase IV CR. The questionnaires will aim to collect data in both quantitative (1-5 Likert scale style responses) and qualitative forms with questions including demographic and reasons for progressing or not progressing to phase IV CR. A convenience sample will be asked to complete a semi-structured interview over the phone or via Microsoft teams, which will last around 20 minutes.

An initiator will be defined as a participant who has attended at least three phase IV CR sessions, and a non-initiator defined as a participant who is either not going to do any exercise post phase III, or to exercise from home on their own. For this study, we will define phase IV CR as any referral to a long-term structured or unstructured maintenance programme of regular exercise/physical activity organised by a third part

The semi-structured interview approach will include core questions that we ask to each interviewee, flexible probing questions to encourage elaboration, and clarification questions that can be used in instances where a participant's answer is unclear. This semi-structured approach will allow individuals to discuss areas of perceived importance (15) whilst allowing us to collect data that are relevant to the research questions. The interviews will be conducted face-to-face when possible and appropriate or via Microsoft Teams® in situations where logistics or COVID precautions prevent in person discussions. Interviews will be recorded using a Dictaphone or the record function on Microsoft Teams®. Care will be taken to report enough information that allows the findings of the study to resonate with readers while protecting the participants' confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* • Those participating in phase III cardiac rehabilitation and nearing successful completion of the programme

  * Subjects capable of giving informed consent
  * >18 years old
  * Clinically stable
  * Successful completion of an NHS commissioned hospital or community based phase III programme
  * Belong to one of the groups being investigated: Underrepresented groups based on the NACR report, i.e. females and ethnic minorities (defined as all people except those in the "White" ethnic group in Great Britain) (22)

Exclusion Criteria:

* • Unstable/uncontrolled coronary heart disease

  * Those presenting with any significant comorbidities or contraindications to exercise testing or training in accordance with the American College of Sports Medicine (11)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All of those participating in phase III cardiac rehabilitation from underepresented populations
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Questionnaires | These will be distributed to participants approximately 2 weeks after Informed consent is obtained
  The questionnaires issued to all participants, these will collect qualitative and quantitative data.

SECONDARY OUTCOMES:
Semi-structured interviews | Within 2 weeks of return of the individual particiant's questionnaire response
  These will be informal conversations conducted in approximately 1/3 of all participants

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Aneurin Bevan University Hospital, Caerleon, Gwent
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Stockport NHS Foundation Trust, Stockport

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other researchers outside of this project.

REFERENCES:
- [Background] BHF. UK statistics 2021.
- [Background] Dibben G, Faulkner J, Oldridge N, Rees K, Thompson DR, Zwisler AD, Taylor RS. Exercise-based cardiac rehabilitation for coronary heart disease. Cochrane Database Syst Rev. 2021 Nov 6;11(11):CD001800. doi: 10.1002/14651858.CD001800.pub4. PMID 34741536
- [Background] Thomas RJ, King M, Lui K, Oldridge N, Pina IL, Spertus J; American Association of Cardiovascular and Pulmonary Rehabilitation/American College of Cardiology/American Heart Association Cardiac Rehabilitation/Secondary Prevention Performance Measures Writing Committee. AACVPR/ACC/AHA 2007 performance measures on cardiac rehabilitation for referral to and delivery of cardiac rehabilitation/secondary prevention services. Circulation. 2007 Oct 2;116(14):1611-42. doi: 10.1161/CIRCULATIONAHA.107.185734. Epub 2007 Sep 20. No abstract available. PMID 17885210
- [Background] Thomas RJ, King M, Lui K, Oldridge N, Pina IL, Spertus J, Bonow RO, Estes NA 3rd, Goff DC, Grady KL, Hiniker AR, Masoudi FA, Radford MJ, Rumsfeld JS, Whitman GR; AACVPR; ACC; AHA; American College of Chest Physicians; American College of Sports Medicine; American Physical Therapy Association; Canadian Association of Cardiac Rehabilitation; European Association for Cardiovascular Prevention and Rehabilitation; Inter-American Heart Foundation; National Association of Clinical Nurse Specialists; Preventive Cardiovascular Nurses Association; Society of Thoracic Surgeons. AACVPR/ACC/AHA 2007 performance measures on cardiac rehabilitation for referral to and delivery of cardiac rehabilitation/secondary prevention services endorsed by the American College of Chest Physicians, American College of Sports Medicine, American Physical Therapy Association, Canadian Association of Cardiac Rehabilitation, European Association for Cardiovascular Prevention and Rehabilitation, Inter-American Heart Foundation, National Association of Clinical Nurse Specialists, Preventive Cardiovascular Nurses Association, and the Society of Thoracic Surgeons. J Am Coll Cardiol. 2007 Oct 2;50(14):1400-33. doi: 10.1016/j.jacc.2007.04.033. No abstract available. PMID 17903645
- [Background] Squires RW, Montero-Gomez A, Allison TG, Thomas RJ. Long-term disease management of patients with coronary disease by cardiac rehabilitation program staff. J Cardiopulm Rehabil Prev. 2008 May-Jun;28(3):180-6; quiz 187-8. doi: 10.1097/01.HCR.0000320068.35728.12. PMID 18496316
- [Background] Sandercock G, Hurtado V, Cardoso F. Changes in cardiorespiratory fitness in cardiac rehabilitation patients: a meta-analysis. Int J Cardiol. 2013 Aug 10;167(3):894-902. doi: 10.1016/j.ijcard.2011.11.068. Epub 2011 Dec 27. PMID 22206636
- [Background] Taylor C, Tsakirides C, Moxon J, Moxon JW, Dudfield M, Witte K, Ingle L, Carroll S. Exercise dose and all-cause mortality within extended cardiac rehabilitation: a cohort study. Open Heart. 2017 Jul 28;4(2):e000623. doi: 10.1136/openhrt-2017-000623. eCollection 2017. PMID 28878950
- [Background] NACR. Quality and Outcomes Report 2019.
- [Background] Ozemek C, Squires RW. Enrollment and Adherence to Early Outpatient and Maintenance Cardiac Rehabilitation Programs. J Cardiopulm Rehabil Prev. 2021 Nov 1;41(6):367-374. doi: 10.1097/HCR.0000000000000645. PMID 34727555
- [Background] Brawner CA, Girdano D, Ehrman JK, Keteyian SJ. Association Between Phase 3 Cardiac Rehabilitation and Clinical Events. J Cardiopulm Rehabil Prev. 2017 Mar;37(2):111-118. doi: 10.1097/HCR.0000000000000201. PMID 27676465
- [Background] Dohnke B, Nowossadeck E, Muller-Fahrnow W. Motivation and participation in a phase III cardiac rehabilitation programme: an application of the health action process approach. Res Sports Med. 2010 Oct;18(4):219-35. doi: 10.1080/15438627.2010.510032. PMID 21058208
- [Background] American College of Sports Medicine. (2022). Guidelines for Exercise Testing and Prescription (G. Ligouri, Ed.; Eleventh). Wolters Kluwer.
- [Background] Beswick AD, Rees K, Griebsch I, Taylor FC, Burke M, West RR, Victory J, Brown J, Taylor RS, Ebrahim S. Provision, uptake and cost of cardiac rehabilitation programmes: improving services to under-represented groups. Health Technol Assess. 2004 Oct;8(41):iii-iv, ix-x, 1-152. doi: 10.3310/hta8410. PMID 15461879
- [Background] Karmali KN, Davies P, Taylor F, Beswick A, Martin N, Ebrahim S. Promoting patient uptake and adherence in cardiac rehabilitation. Cochrane Database Syst Rev. 2014 Jun 25;(6):CD007131. doi: 10.1002/14651858.CD007131.pub3. PMID 24963623
- [Background] Herber OR, Bucker B, Metzendorf MI, Barroso J. A qualitative meta-summary using Sandelowski and Barroso's method for integrating qualitative research to explore barriers and facilitators to self-care in heart failure patients. Eur J Cardiovasc Nurs. 2017 Dec;16(8):662-677. doi: 10.1177/1474515117711007. Epub 2017 May 16. PMID 28509565
- [Background] Sparkes, A. C., & Smith, B. (2014). Qualitative research methods in sport, exercise and health: From process to product. Routledge/Taylor & Francis Group.
- [Background] QSR International Pty Ltd. (2020) NVivo (released in March 2020), https://www.qsrinternational.com/nvivo-qualitative-data-analysis-software/home
- [Background] Braun V, Clarke V. Novel insights into patients' life-worlds: the value of qualitative research. Lancet Psychiatry. 2019 Sep;6(9):720-721. doi: 10.1016/S2215-0366(19)30296-2. Epub 2019 Jul 23. No abstract available. PMID 31350207
- [Background] Merriam, S. B., & Tisdell, E. J. (2016). Qualitative Research: A Guide to Design and Implementation (4th ed.). San Francisco, CA: Jossey Bass.
- [Background] Denzin, N. K. (1978). Triangulation: A Case for Methodological Evaluation and Combination. Sociological Methods, 339-357.
- [Background] Patton, M. Q. (2015). Qualitative research and evaluation methods: Theory and practice; Fourth Edition. In SAGE Publications, Inc.
- [Background] Ethnic diversity in politics and public life - House of Commons Library. (n.d.). Retrieved October 10, 2022, from https://commonslibrary.parliament.uk/research-briefings/sn01156/
- [Background] Ryba, T. V., Haapanen, S., Mosek, S., & Ng, K. (2012). Toward a conceptual understanding of acute cultural adaptation: A preliminary examination of ACA in female swimming. Qualitative Research in Sport, Exercise and Health, 4(1), 80-97. https://doi.org/10.1080/2159676X.2011.653498